CLINICAL TRIAL: NCT06668090
Title: Biochemical Bone Turnover Markers and Bone Mechanical Properties Following Exercise Induced Changes in Insulin Sensitivity in People With Type 2 Diabetes
Brief Title: Bone Properties Following Exercise Induced Changes in Insulin Sensitivity in People With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: The Novo Nordic Foundation (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Søren Gregersen, Clinical Associate Professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-221-19
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance; Bone Diseases, Metabolic; Osteoporosis, Osteopenia; Musculoskeletal Diseases; Metabolic Disease; Glucose Metabolism Disorders
Keywords: Diabetes Mellitus, Type 2; Bone; Bioelectric impedance; Diabetic bone disease; Insulin supression test (IST); Bone turnover
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Bone Diseases, Metabolic; Osteoporosis; Musculoskeletal Diseases; Metabolic Diseases; Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental): Moderate intensity bike exercise thrice weekly for 12 week added to the usual activity level.
  Each participant receive an individual exercise program based on their maximum heart rate.
  Exercise is not supervised, but compliance is monitored. It will either be performed at home or at gyms.
  No changes in diet.
  Interventions: Behavioral: Moderate intensity bike exercise
- Control/no intervention (No Intervention): 12 weeks with usual activity level.
  No changes in diet.

INTERVENTIONS:
Behavioral: Moderate intensity bike exercise — Participants will do moderate intensity bike exercise for up to one hour thrice weekly for 12 weeks.
  Arms: Exercise

SUMMARY:
Diabetes mellitus type 2 is associated with low bone turnover and increased risk of bone fractures.

Bone mineral density, however, is increased and cannot explain the increased fracture risk per se. The pathophysiology is not completely understood, but the decrease in bone turnover is believed to cause an accumulation of microcracks in bone tissue leading to bone fragility. The decrease in bone turnover may arise directly from insulin resistance or indirectly through formation of advanced glycation end-products.

The main aim objective is to investigate how increases in insulin sensitivity following 12 weeks of moderate intensity bike exercise affect biochemical bone turnover markers and biomechanical bone properties in individuals with diabetes mellitus type 2.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 2
* Age ≥ 45 years
* Male or female sex
* Women must be postmenopausal

Exclusion Criteria:

* Recent substantial changes in diet (within 3 months)
* Recent substantial changes in activity level (within 3 months)
* Recent substantial weight changes (within 3 months)
* Current or previous treatment (within the last 2 years) with non-oral anti-diabetics or oral GLP-1 analogs
* HbA1c ≥ 90 mmol/mol
* HbA1c < 48 mmol/mol without anti-diabetic medication
* Premature menopause (menopause before 40 years of age)
* Current pregnancy
* Treatment with one of the following medications:

  * Systemic glucocorticoids (within the last 2 years)
  * Antiresorptive or bone anabolic medication (ever)
  * Lithium (ever)
  * Anticonvulsive medication (current)
  * Menopausal replacement therapy (currently)
* Estimered glomerular filtrationsrate (eGFR) < 60 mL/minutes
* High level of physical activity, assessed by the investigators to interfere with the study results
* Substantial cardiovascular, endocrine, renal, hepatic, rheumatological, gastrointestinal or other disorders assessed by the investigator
* Electronic implants
* Osteoporosis or other bone disease
* Resent bone fracture (within 6 months)
* Previous bone fracture in either both tibial bones or both radial bones
* Parathyroid or calcium metabolism disorder
* Vitamin D deficiency (< 50 nmol/L)
* Other substantial medical disorder in unstable phase or active cancer within the last five years except spino- or basocellular carcinoma
* Lack of ability to complete the intervention
* Patients assessed uneligible by the investigator to participate in the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-28 (Actual)

PRIMARY OUTCOMES:
Steady state plasma glucose during stage 1 of insulin suppression test (mmol/L) | 100, 110 and 120 minutes after test-start. 12-week change. Comparison between pre-intervention and end-intervention steady state plasma glucose.
  Subjects are administered a 25 μg octreotide bolus at time-point 0 minutes and subsequently infused with 0.27 μg octreotide / m2 • minute, 6 milliunits (mU) insulin / m2 • minute, and 50 mg glucose / m2 • min.
Steady state plasma glucose during stage 2 of insulin suppression test (mmol/L) | 220, 230 and 240 minutes after test-start. 12-week change. Comparison between pre-intervention and end-intervention steady state plasma glucose
  Subjects are administered a 25 μg octreotide bolus at time-point 0 minutes and subsequently infused with 0.27 μg octreotide / m2 • minute, 6 (mU) insulin / m2 • minute, and 50 mg glucose / m2 • minute. At time-point 120 minutes, infusion speeds are increased to to 32 mU insulin / m2 • minute and 267 mg glucose / m2 • minute.

SECONDARY OUTCOMES:
Hemoglobin A1c (mmol/mol) | 12-week change. Comparison between pre-intervention and end-intervention
  During fasting.
Fasting Homeostatic Model Assessment for Insulin Resistance by C-peptide (arbitrary unit). | 12-week change. Comparison between pre-intervention blood samples and end-intervention blood samples.
Circulating glucose (mmol/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Circulating insulin (pmol/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Alkaline phosphatase (total and bone type) (U/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Circulating CTX (µg/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Measured during fasting and during stage 1 and 2 of the insulin suppression test They are measured during fasting and during stage 1 and 2 of the insulin suppression test
Circulating Osteocalcin (µg/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Measured during fasting and during stage 1 and 2 of the insulin suppression test
Circulating Osteoglycin (µg/l) | 12-week change. Comparison between pre-intervention and end-intervention
  They are measured during fasting and during stage 1 and 2 of the insulin suppression test
Circulating P1NP (µg/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Measured during fasting and during stage 1 and 2 of the insulin suppression test
Circulating Sclerostin (µg/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Measured during fasting and during stage 1 and 2 of the insulin suppression test
Ionized calcium (mmol/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Circulating Parathyroid hormone (pmol/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Measured during fasting and during stage 1 and 2 of the insulin suppression test
Vitamin D (nmol/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Bone Mineral Density (t-score) in hip and spine | 12-week change. Comparison between pre-intervention and end-intervention
  Dual-energy X-ray absorptiometry (DXA).
Advanced glycation end-products (AGEs) in skin | 12-week change. Comparison between pre-intervention and end-intervention
  Measurement of skin autofluorescence in the forearm
Results from the HRpQCT scan including trabecular and cortical state | 12-week change. Comparison between pre-intervention and end-intervention
  Measured in the tibial and radial bone on the non-dominant side
Body composition assessed with whole-body Dual-energy X-ray absorptiometry (DXA) | 12-week change. Comparison between pre-intervention and end-intervention
  Measured during fasting
FIB-4 score | 12-week change. Comparison between pre-intervention and end-intervention
  Using age, ALAT, ASAT and thrombocytes
Alanine aminotransferase (unit(U)/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Aspartate aminotransferase (U)/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Thrombocytes (10^9/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Bioelectric impedance analysis (BIA) | 12-week change. Comparison between pre-intervention and end-intervention
  Following measurements will be evaluated: Phase angle, membrane capacitance, impedance, capacitive resistance, resistance.
  Measured during fasting and stage 1 and 2 of insulin suppression test
Steady state glycerol and free fatty acids during stage 1 and 2 of insulin suppression test (mmol/L) | 100, 110, 120, 220, 230 and 240 minutes after test-start. 12-week change. Comparison between pre-intervention and end-intervention steady state plasma glucose.
  Subjects are administered a 25 μg octreotide bolus at time-point 0 minutes and subsequently infused with 0.27 μg octreotide / m2 • minute, 6 (mU) insulin / m2 • minute, and 50 mg glucose / m2 • minute. At time-point 120 minutes, infusion speeds are increased to to 32 mU insulin / m2 • minute and 267 mg glucose / m2 • minute.
Total cholesterol (mmol/l), | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Low density lipoprotein (LDL) (mmol/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
High density lipoprotein (HDL) (mmol/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Fastomg
Triglycerides (mmol/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Blood pressure (mmHg) | 12-week change. Comparison between pre-intervention and end-intervention
  Average daytime and night-time ambulatory blood pressure. 24-hour ambulatory blood pressure measurement, measured every 20 minutes during daytime and every 30 minutes during nighttime.
Body composition assessed with bioelectric impedance analysis (BIA) | 12-week change. Comparison between pre-intervention and end-intervention
  Measured during fasting
Circulating adiponectin | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Leptin (n/mL) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Alpha-hydroxybutyrate (μg/mL) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Monocyte chemoattractant protein-1 (pg/ml) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Interleukin 1 beta (pg/ml) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Interleukin 6 (pg/ml) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Estimated glomerular filtration rate (ml/min/1,73m2) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting

OTHER OUTCOMES:
Thyroid-stimulating hormone (international unit (IU)/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
High sensitivity C reactive protein (mg/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Thyroid stimulating hormone (pmol/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Creatinine (μmol/l) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting
Activity tracking | 12-week change. Comparison between pre-intervention and end-intervention
  Measured with accelerometer on thigh of non-dominant leg
Activity level - questionnaire | 12-week change. Comparison between pre-intervention and end-intervention
Diet diary (3 days) | 12-week change. Comparison between pre-intervention and end-intervention
Urine albumin-to-creatinine ratio (mg/g) | 12-week change. Comparison between pre-intervention and end-intervention
  Fasting

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus N, Denmark